CLINICAL TRIAL: NCT05169021
Title: Folic Acid and Intensive Antihypertensive Therapy for Cerebrovascular and Cardiovascular Events Prevention Among Patients With Hypertension and Cerebral Small Vascular Diseases (FAITH)----A Multicenter, Randomized, Controlled, Open-label, 2x2 Factorial, Blinded End-point Trial
Brief Title: Folic Acid and Intensive Antihypertensive Therapy for Hypertension With CSVD
Acronym: FAITH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, President of Beijing Tiantan Hospital, Capital Medical University, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAITH
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Cerebral Small Vessel Diseases; Stroke
Keywords: Cerebral Small Vessel Diseases; Stroke recurrence; Hypertension; Homocysteine; Folic acid
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Stroke; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amlodipine folic acid 5.8mg+intensive antihypertensive therapy (Active Comparator): This group will receive intensive antihypertensive therapy (systolic blood pressure(SBP) <130 mmHg); with amlodipine folic acid 5.8mg.
  Interventions: Drug: Amlodipine folic acid 5.8mg+intensive antihypertensive therapy
- Amlodipine folic acid 5.8mg+standard antihypertensive therapy (Active Comparator): This group will receive standard antihypertensive therapy (SBP: 130-140 mmHg); with amlodipine folic acid 5.8mg.
  Interventions: Drug: Amlodipine folic acid 5.8mg+standard antihypertensive therapy
- Amlodipine+intensive antihypertensive therapy (Active Comparator): This group will receive intensive antihypertensive therapy (systolic blood pressure(SBP) <130 mmHg); with amlodipine 5.0mg.
  Interventions: Drug: Amlodipine+intensive antihypertensive therapy
- Amlodipine+standard antihypertensive therapy (Placebo Comparator): This group will receive standard antihypertensive therapy (SBP: 130-140 mmHg); with amlodipine 5.0mg.
  Interventions: Drug: Amlodipine+standard antihypertensive therapy

INTERVENTIONS:
Drug: Amlodipine folic acid 5.8mg+intensive antihypertensive therapy — Amlodipine folic acid tablet 5.8mg, taken daily, in the morning after waking.
  To achieve target blood pressure(SBP<130mmHg), this study will provide, if needed, concurrent antihypertensive medications. Patients will be asked to discontinue all prior concurrent medications. Recommended treatment options are described below:
  1. Add candesartan 4mg;
  2. Add indapamide 2.5mg;
  3. Increase dose of candesartan to 8mg;
  4. Increase dose of amlodipine to 7.5mg-10mg.
  Arms: Amlodipine folic acid 5.8mg+intensive antihypertensive therapy
Drug: Amlodipine folic acid 5.8mg+standard antihypertensive therapy — Amlodipine folic acid tablet 5.8mg, taken daily, in the morning after waking.
  To achieve target blood pressure (SBP:130-140mmHg), this study will provide, if needed, concurrent antihypertensive medications. Patients will be asked to discontinue all prior concurrent medications. Recommended treatment options are described below:
  1. Add candesartan 4mg;
  2. Add indapamide 2.5mg;
  3. Increase dose of candesartan to 8mg;
  4. Increase dose of amlodipine to 7.5mg-10mg.
  Arms: Amlodipine folic acid 5.8mg+standard antihypertensive therapy
Drug: Amlodipine+intensive antihypertensive therapy — Amlodipine tablet 5.8mg, taken daily, in the morning after waking.
  To achieve target blood pressure (SBP: 130-140 mmHg), this study will provide, if needed, concurrent antihypertensive medications. Patients will be asked to discontinue all prior concurrent medications. Recommended treatment options are described below:
  1. Add candesartan 4mg;
  2. Add indapamide 2.5mg;
  3. Increase dose of candesartan to 8mg;
  4. Increase dose of amlodipine to 7.5mg-10mg.
  Arms: Amlodipine+intensive antihypertensive therapy
Drug: Amlodipine+standard antihypertensive therapy — Amlodipine tablet 5.8mg, taken daily, in the morning after waking.
  To achieve target blood pressure (SBP: 130-140 mmHg), this study will provide, if needed, concurrent antihypertensive medications. Patients will be asked to discontinue all prior concurrent medications. Recommended treatment options are described below:
  1. Add candesartan 4mg;
  2. Add indapamide 2.5mg;
  3. Increase dose of candesartan to 8mg;
  4. Increase dose of amlodipine to 7.5mg-10mg.
  Other Names: Standard antihypertensive therapy
  Arms: Amlodipine+standard antihypertensive therapy

SUMMARY:
The primary objectives of this trial are:

1. Efficacy evaluation of amlodipine folic acid tablets:

   To assess the effects of amlodipine folic acid tablets 5.8 mg (5 mg amlodipine + 0.8 mg folic acid)versus amlodipine tablets 5 mg in preventing all-cause stroke in cerebral small vascular disease (CSVD) patients with hypertension and elevated homocysteine (Hcy) level.
2. Intensive Antihypertensive Therapy:

To assess the effect of intensive antihypertensive therapy (SBP<130 mmHg) versus standard antihypertensive therapy (SBP 130-<140 mmHg) in reducing risk of combined cardio-cerebrovascular events in CSVD patients with hypertension and elevated Hcy level, using two basic anti-hypertensive drugs, amlodipine tablets 5 mg or amlodipine folic acid tablets 5.8 mg.

DETAILED DESCRIPTION:
Hypertension is highly prevalent risk factor for stroke, particularly for stroke associated with CSVD. Blood pressure (BP) lowering has been considered an important measure for preventing stroke and progression of CSVD. Moreover, uncertainty remains regarding the efficacy of folic acid therapy for secondary prevention of stroke because of limited and inconsistent data. We propose to conduct a randomized, double-blind, placebo-controlled, multicenter, 2×2 factorial designed clinical trial to test the primary hypothesis that 1) whether amlodipine folic acid is more effective than amlodipine in reducing the risk of all-cause stroke (including fatal and non-fatal stroke) over a follow-up period among patients with CSVD. 2) whether an intensive treatment strategy (a systolic BP target of <130mmHg) is more effective than a standard treatment strategy (a systolic BP target of 130-140mmHg) in reducing the risk of combined cardio-cerebrovascular events.

Both Intention-to-treat Analysis (ITT) and Per-protocol set (PPS) were used for analysis.

We will use Kaplan-Meier estimates of the cumulative risk of stroke (ischemic or hemorrhagic) event and combined cardio-cerebrovascular events during follow-up period, with hazards ratios and 95% CI calculated using Cox proportional hazards methods and the log-rank test to evaluate the treatment effect. All statistics will be 2-sided with P<0.05 considered significant, accounting for interim analyses.

All patients who received study drugs and with at least one safety follow-up record will be included in the safety population. The data for safety evaluation included adverse reactions observed during the trial and changes in laboratory data before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-75 years;
2. Meets any of the following criteria:

1) Lacunar infarction occurring within the period of seven days up to one year post-infarction, diagnosed by head MRI/CT (meeting modified Fisher criteria*); 2）Head MRI indicating white matter hyperintensity, 4≥Fazekas score*≥2; 3）Head MRI indicating white matter hyperintensity, Fazekas=1, combined with old subcortical vascular lacunar infarction;

* For modified Fisher criteria and Fazekas score, see FAITH main study appendix 1 and appendix 6).

  3. Medical recorded history of hypertension. Systolic blood pressure SBP: 130-180 mm Hg on 0 or 1 medication SBP: 130-170 mm Hg on up to 2 medications SBP: 130-160 mm Hg on up to 3 medications. 4. mRS score ≤2; 5. Serum Hcy ≥10 µmol/L or MTHFR 677 TT genotype; 6. Signed informed consent form.

Exclusion Criteria:

1. Patients with secondary hypertension;
2. Symptomatic intracranial and extracranial artery stenosis (stenosis ≥50%), or asymptomatic intracranial and extracranial artery stenosis (stenosis≥70%);
3. Patients who have undergone revascularization of the heart, brain, or kidney, or other aortic stenting procedures;
4. Any symptoms of orthostatic hypotension when measuring standing blood pressure, or if standing SBP <110mmHg;
5. Bilateral renal artery stenosis;
6. Patients who have previously taken candesartan or other angiotensin receptor antagonist (ARB) type medication, indapamide or other similar diuretic type medication, or any medication or health product containing folic acid, and reported adverse reactions;
7. Patients who have indicators for specific antihypertensive medications (e.g. β-blockers after acute myocardial infarction, RAS blockers for prevention of cardiovascular disease, α-blockers for treatment of benign prostate hyperplasia);
8. Within the last three months, regular usage of vitamin supplements containing folic acid, B6, or B12, or usage of folic acid antagonists (e.g. methotrexate);
9. Patients undergoing dialysis or with stage 4-5 chronic kidney disease, or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m²;
10. History of epilepsy or currently using anti-epileptic medication;
11. Pregnant and lactating women, or women planning to become pregnant;
12. Life expectancy less than four years;
13. Within the last month, participation in another clinical trial;
14. Any patient determined by the researchers to be unsuitable for the present study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause stroke (including fatal and non-fatal stroke) | 4 year after randomization
  This aims to assess the effects of amlodipine folic acid tablets 5.8 mg (5 mg amlodipine + 0.8 mg folic acid)versus amlodipine tablets 5 mg in preventing stroke occurrence in cerebral small vascular disease (CSVD) patients with hypertension and elevated homocysteine (Hcy) level
Combined cardio-cerebrovascular events | 4 year after randomization
  This aims to assess the effect of intensive antihypertensive therapy (SBP<130 mmHg) versus standard antihypertensive therapy (SBP 130-<140 mmHg) in reducing risk of combined cardio-cerebrovascular events in CSVD patients with hypertension and elevated Hcy level.

SECONDARY OUTCOMES:
Combined cardio-cerebrovascular events | 4 year after randomization
  Secondary outcome for assessing the effects of amlodipine folic acid tablets 5.8 mg (5 mg amlodipine + 0.8 mg folic acid)versus amlodipine tablets 5 mg in preventing combined cardio-cerebrovascular events in cerebral small vascular disease (CSVD) patients with hypertension and elevated homocysteine (Hcy) level.
All-cause stroke (including fatal and non-fatal stroke) | 4 year after randomization
  Secondary outcome for assessing the effect of intensive antihypertensive therapy (SBP<130 mmHg) versus standard antihypertensive therapy (SBP 130-<140 mmHg) in reducing risk of stroke occurrence in CSVD patients with hypertension and elevated Hcy level.
Ischemic stroke | 4 year after randomization
  Percentage of patients within follow-up period new ischemic stroke events.
Hemorrhagic stroke | 4 year after randomization
  Percentage of patients within follow-up period new hemorrhagic stroke events.
Myocardial infarction | 4 year after randomization
  Percentage of patients within follow-up period new myocardial infarction events.
Hospitalization from heart failure | 4 year after randomization
  Hospitalization, or an emergency department visit requiring treatment with infusion therapy, for a clinical syndrome that presents with multiple signs and symptoms consistent with cardiac decompensation/ inadequate cardiac pump function within follow-up period.
Cardio-cerebrovascular death | 4 year after randomization
  Cardio-cerebrovascular death includes death caused by acute myocardial infarction (MI), sudden cardiac death, death caused by heart failure (HF), death caused by stroke, death caused by cardiovascular surgery, death caused by cardiovascular hemorrhage and other cardiovascular causes.
All-cause death | 4 year after randomization
  This is death due to various causes, including cardiovascular and non-vascular deaths and deaths from unknown causes.

OTHER OUTCOMES:
Malignant tumors occurence | 4 year after randomization
  To assess the effects of amlodipine folic acid tablets 5.8 mg (5 mg amlodipine + 0.8 mg folic acid)versus amlodipine tablets 5 mg in preventing malignant tumors occurrence in cerebral small vascular disease (CSVD) patients with hypertension and elevated homocysteine (Hcy) level.
Changes in total image load score of CSVD | 4 year after randomization
  Changes in total image load score of CSVD
Changes in WMLs and brain volume | 4 year after randomization
  Changes in WMLs and brain volume
Changes in score of each single item of the grading of CSVD image load | 4 year after randomization
  Changes in score of each single item of the grading of CSVD image load
Changes in autonomic nervous system function and cerebral hemodynamics | 4 year after randomization
  Changes in autonomic nervous system function and cerebral hemodynamics
Changes in MoCA score | 4 year after randomization
  Changes in MoCA score

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huo Y, Li J, Qin X, Huang Y, Wang X, Gottesman RF, Tang G, Wang B, Chen D, He M, Fu J, Cai Y, Shi X, Zhang Y, Cui Y, Sun N, Li X, Cheng X, Wang J, Yang X, Yang T, Xiao C, Zhao G, Dong Q, Zhu D, Wang X, Ge J, Zhao L, Hu D, Liu L, Hou FF; CSPPT Investigators. Efficacy of folic acid therapy in primary prevention of stroke among adults with hypertension in China: the CSPPT randomized clinical trial. JAMA. 2015 Apr 7;313(13):1325-35. doi: 10.1001/jama.2015.2274. PMID 25771069
- [Result] Toole JF, Malinow MR, Chambless LE, Spence JD, Pettigrew LC, Howard VJ, Sides EG, Wang CH, Stampfer M. Lowering homocysteine in patients with ischemic stroke to prevent recurrent stroke, myocardial infarction, and death: the Vitamin Intervention for Stroke Prevention (VISP) randomized controlled trial. JAMA. 2004 Feb 4;291(5):565-75. doi: 10.1001/jama.291.5.565. PMID 14762035
- [Result] VITATOPS Trial Study Group. B vitamins in patients with recent transient ischaemic attack or stroke in the VITAmins TO Prevent Stroke (VITATOPS) trial: a randomised, double-blind, parallel, placebo-controlled trial. Lancet Neurol. 2010 Sep;9(9):855-65. doi: 10.1016/S1474-4422(10)70187-3. Epub 2010 Aug 3. PMID 20688574
- [Result] SPS3 Study Group; Benavente OR, Coffey CS, Conwit R, Hart RG, McClure LA, Pearce LA, Pergola PE, Szychowski JM. Blood-pressure targets in patients with recent lacunar stroke: the SPS3 randomised trial. Lancet. 2013 Aug 10;382(9891):507-15. doi: 10.1016/S0140-6736(13)60852-1. Epub 2013 May 29. PMID 23726159
- [Result] Croall ID, Tozer DJ, Moynihan B, Khan U, O'Brien JT, Morris RG, Cambridge VC, Barrick TR, Blamire AM, Ford GA, Markus HS; PRESERVE Study Team. Effect of Standard vs Intensive Blood Pressure Control on Cerebral Blood Flow in Small Vessel Disease: The PRESERVE Randomized Clinical Trial. JAMA Neurol. 2018 Jun 1;75(6):720-727. doi: 10.1001/jamaneurol.2017.5153. PMID 29507944